CLINICAL TRIAL: NCT00737711
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Two Weekly Administration of Intravenous Methoxy Polyethylene Glycol-epoetin Beta (MIRCERA) for the Treatment of Chronic Renal Anemia in Dialysis Patients Not Currently Treated With Erythropoietin-stimulating Agent (ESA).
Brief Title: A Study of Two-Weekly Intravenous Mircera for the Treatment of Dialysis Patients With Chronic Renal Anemia Not Receiving ESA Therapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21822
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — iv 0.6 micrograms/kg every 2 weeks

SUMMARY:
This single arm study will evaluate the hemoglobin (Hb) increasing effect, safety and tolerability of two-weekly intravenous administration of Mircera in dialysis patients with chronic renal anemia not currently treated with ESAs. Patients will receive intravenous Mircera 0.6 micrograms/kg every 2 weeks for 16 weeks with follow up 2 weeks after the last treatment visit. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, >=18 years of age;
* chronic renal anemia (Hb concentration 8.0g/dL - 10.0g/dL);
* no prior erythropoietin stimulating agent (ESA) therapy.

Exclusion Criteria:

* blood transfusion within the previous 4 weeks;
* poorly controlled hypertension;
* significant acute or chronic bleeding;
* active malignant disease;
* congestive heart failure (NYHA Class IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- India (13):
  - Ahmedabad
  - Bangalore
  - Chennai
  - Coimbatore
  - Gujarat
  - Hyderabad
  - Kerala
  - Kolkata
  - Ludhiana
  - Mumbai
  - New Delhi
  - Vellore
  - Vishakpatnam

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 08 July 2008 to 31 May 2009 across 16 centers in India. A total of 189 participants were enrolled in the study.
Groups:
- MIRCERA: Participants with chronic renal anemia, on dialysis, received 0.6 microgram per kilogram of body weight (mcg/kg) of Methoxy polyethylene glycol-epoetin beta (MIRCERA/RO0503821), intravenously once every two weeks for 16 weeks. A telephonic / physical follow-up visit took place 2 weeks after the end of the MIRCERA treatment period.
Period: Overall Study
Arm/Group | MIRCERA
Started | 189
Completed | 158
Not Completed | 31
Not completed — Adverse Event | 2
Not completed — Death | 8
Not completed — Failure to return | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Blood transfusion | 6
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who receive at least one dose of study medication.
Groups:
- MIRCERA: Participants with chronic renal anemia, on dialysis, received 0.6 mcg/kg MIRCERA, intravenously once every two weeks for 16 weeks. A telephonic or physical follow-up visit took place 2 weeks after the end of the MIRCERA treatment period.
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.74 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 139

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Concentration From Baseline to Week 16 of the Treatment Period
Description: The difference between the mean Hemoglobin (Hb) value at the last visit (Week 16) of the treatment period (TP) and at Baseline (Week 0) is presented. TP was from Baseline to Week 16.
Time Frame: Baseline (Week 0) and Week 16
Population: The intent-to-treat (ITT) population included all participants who received at least one dose of the study drug. Data for participants available at the time of assessment is presented.
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dL)
Arm/Group | MIRCERA
Number analyzed (Participants) | 159
gram/deciliter (g/dL) | 2.11 (1.30)
Statistical Analysis 1: Comparison: MIRCERA; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test was used to estimation of p-value

2. Secondary Outcome: Mean Time Required to Achieve Blood Hemoglobin Levels Within Target Range of 10.0-12.0 Gram/Deciliter
Description: Achievement of blood Hb levels within target range of 10.0-12.0 g/dL was considered as achievement of response. The mean time required to achieve the Hb target range is presented in weeks.
Time Frame: Up to Week 16
Population: The ITT population included all participants who received at least one dose of the study drug. Data for participants available at the time of assessment is presented.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | MIRCERA
Number analyzed (Participants) | 144
Weeks | 6.10 (3.87)

3. Secondary Outcome: Mean Time Spent in the Hemoglobin Range of 10.0-12.0 Gram/Deciliter From Week 12 to Week 16
Description: The Hb concentration was recorded for all the participants at enrollment and different time points throughout the study up to Week 16. The mean time spent (in weeks) by the participants in the target range (10-12 g/dL) during the last 4 weeks of the TP is presented.
Time Frame: Week 12 to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | MIRCERA
Number analyzed (Participants) | 103
Weeks | 3.07 (1.00)

4. Secondary Outcome: Percentage of Participants With Average Hemoglobin Concentration Between 10.0-12.0 Gram/Deciliter From Week 12 to Week 16
Description: The Hb concentration was recorded for all the participants at enrollment and different time points throughout the study up to Week 16. The percentage of participants achieving Hb levels within target range of 10.0-12.0 g/dL during the last 4 weeks of the TP is presented.
Time Frame: Week 12 to Week 16
Population: The ITT population included all participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
percentage of participants | 46.20 [38.56 to 53.97]

5. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths
Description: An adverse event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. A serious adverse event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution. An SAE is any AE that can result in death or is life-threatening or required participant hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect; or is medically significant or requires intervention to prevent one or other of the outcomes listed above
Time Frame: Up to Week 18
Population: Safety population included all participants who receive at least one dose of study drug, and for whom all safety parameters were listed in individual participant listings, by visit, center and participant number.
Measure: Number; unit: Participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
Participants
  Participants with any AE | 53
  Participants with SAE | 24
  Deaths | 8

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram
Description: Twelve-lead electrocardiogram (ECG) was recorded for the participants. The number of participants with abnormal ECG is presented.
Time Frame: Up to Week 16
Population: Safety population included all participants who receive at least one dose of study drug, and for whom all safety parameters were listed in individual participant listings, by visit, center and participant number. n = the number of participants analyzed at a given time point.
Measure: Number; unit: Participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
Participants
  Participants with abnormal ECG, Week 0, n=189 | 52
  Participants with abnormal ECG, Week 16, n=164 | 49

7. Secondary Outcome: Number of Participants With Reports of Blood Transfusions
Description: Indications for blood transfusions were acute blood loss (bleeding), lack of treatment response or treatment failure, or other reasons.
Time Frame: Up to Week 16
Population: The ITT population included all participants who receive at least one dose of study drug. Participants available at the time of assessment were included.
Measure: Number; unit: Participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
Participants
  White blood cells transfusions | 1
  Pack cell transfusions | 6
  Pure red cell transfusions | 0

8. Secondary Outcome: Number of Participants With Reports of Anti-Epoetin Antibodies
Description: Participants were assessed for the presence of Anti-Epoetin antibodies for MIRCERA.
Time Frame: Up to Week 16
Population: The ITT population included all participants who receive at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 189
Participants | 0

9. Secondary Outcome: Mean White Blood Cell Count Over Time
Description: The mean values of white blood cells are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | MIRCERA
Number analyzed (Participants) | 187
cells per cubic millimeter
  Week 0, n = 187 | 9382.89 (11644.69)
  Week 4, n = 173 | 9181.27 (12689.96)
  Week 10, n = 167 | 9361.38 (13319.73)
  Week 16, n = 159 | 9023.71 (13109.61)

10. Secondary Outcome: Mean Value of Mean Corpuscular Volume Over Time
Description: Mean corpuscular volume (MCV) is a measure of the average volume of red blood corpuscles (RBCs) and is calculated by dividing hematocrit value by the concentration of RBCs. Mean values of MCV are presented at Baseline (Week 0), Week 4, Week 10, and Week 16. Reference range of mean corpuscular volume is 80-96 femtoliter (fL) per red blood cell.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | MIRCERA
Number analyzed (Participants) | 183
Femtoliter
  Week 0, n = 183 | 87.05 (11.37)
  Week 4, n = 169 | 89.17 (6.99)
  Week 10, n = 167 | 88.46 (6.85)
  Week 16, n = 159 | 88.03 (9.36)

11. Secondary Outcome: Mean Hypochromic Red Blood Cells Over Time
Description: Mean values of hypochromic RBCs are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | MIRCERA
Number analyzed (Participants) | 39
cells per cubic millimeter
  Week 0, n = 39 | 3.84 (5.78)
  Week 4, n = 39 | 2.74 (1.13)
  Week 10, n = 36 | 3.23 (1.27)
  Week 16, n = 31 | 3.52 (1.50)

12. Secondary Outcome: Mean Platelet Count Over Time
Description: Mean values of platelet count are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | MIRCERA
Number analyzed (Participants) | 186
cells per cubic millimeter
  Week 0, n = 186 | 214629.03 (77442.90)
  Week 4, n = 177 | 203050.85 (81720.79)
  Week 10, n = 167 | 204922.16 (78064.46)
  Week 16, n = 158 | 194550.63 (78937.74)

13. Secondary Outcome: Mean Serum Iron Over Time
Description: Mean values of serum iron are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram/deciliter (mcg/dL)
Arm/Group | MIRCERA
Number analyzed (Participants) | 187
microgram/deciliter (mcg/dL)
  Week 0, n = 187 | 91.72 (53.44)
  Week 4, n = 171 | 80.17 (39.45)
  Week 10, n = 166 | 87.62 (42.90)
  Week 16, n = 157 | 91.70 (47.36)

14. Secondary Outcome: Mean Serum Ferritin Over Time
Description: Mean values of serum ferritin are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram /milliliter (ng/mL)
Arm/Group | MIRCERA
Number analyzed (Participants) | 188
nanogram /milliliter (ng/mL)
  Week 0, n = 188 | 963.28 (2398.89)
  Week 4, n = 170 | 702.37 (679.50)
  Week 10, n = 161 | 686.42 (723.22)
  Week 16, n = 153 | 641.26 (627.66)

15. Secondary Outcome: Mean Transferrin Over Time
Description: Mean values of serum transferrin are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | MIRCERA
Number analyzed (Participants) | 73
milligram per deciliter (mg/dL)
  Week 0, n = 73 | 173.48 (108.93)
  Week 4, n = 66 | 176.97 (105.16)
  Week 10, n = 55 | 237.98 (304.97)
  Week 16, n = 58 | 181.50 (174.83)

16. Secondary Outcome: Mean Total Iron-binding Capacity Over Time
Description: Mean values of total iron-binding capacity are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 185
mcg/dL
  Week 0, n = 185 | 247.06 (64.08)
  Week 4, n = 166 | 243.25 (71.20)
  Week 10, n = 160 | 245.30 (69.25)
  Week 16, n = 153 | 245.30 (70.03)

17. Secondary Outcome: Mean Transferrin Saturation Over Time
Description: Transferrin saturation (TSAT) measured as a percentage, is a medical laboratory test. It is calculated as serum iron/ total iron-binding capacity x 100. Mean values of transferrin saturation at Baseline (Week 0), Week 4, Week 10, and Week 16 are presented.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of transferrin saturation
Arm/Group | MIRCERA
Number analyzed (Participants) | 186
Percentage of transferrin saturation
  Week 0, n = 186 | 40.39 (27.87)
  Week 4, n=168 | 35.31 (22.46)
  Week 10, n=161 | 36.91 (18.85)
  Week 16, n = 153 | 38.31 (21.27)

18. Secondary Outcome: Mean Serum Albumin Over Time
Description: Mean values of serum albumin are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 185
g/dL
  Week 0, n = 185 | 3.51 (0.54)
  Week 4, n = 172 | 3.48 (0.53)
  Week 10, n = 167 | 3.57 (0.57)
  Week 16, n = 155 | 3.61 (0.54)

19. Secondary Outcome: Mean Serum Globulin Over Time
Description: Mean values of serum globulin are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 179
g/dL
  Week 0, n = 179 | 3.36 (0.67)
  Week 4, n = 163 | 3.24 (0.63)
  Week 10, n = 159 | 3.33 (0.63)
  Week 16, n = 150 | 3.50 (2.50)

20. Secondary Outcome: Mean Serum Creatinine Over Time
Description: Mean values of serum creatinine are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 186
mg/dL
  Week 0, n = 186 | 8.25 (3.05)
  Week 4, n = 171 | 8.65 (3.09)
  Week 10, n = 168 | 9.48 (7.69)
  Week 16, n = 158 | 9.05 (3.31)

21. Secondary Outcome: Mean Blood Urea Nitrogen Over Time
Description: Mean values of blood urea nitrogen (BUN) are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 181
mg/dL
  Week 0, n = 181 | 68.98 (48.61)
  Week 4, n = 170 | 66.19 (42.13)
  Week 10, n = 168 | 67.21 (42.29)
  Week 16, n = 157 | 69.88 (47.77)

22. Secondary Outcome: Mean Serum Potassium Over Time
Description: Mean values of serum potassium are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | MIRCERA
Number analyzed (Participants) | 183
millimoles per liter (mmol/L)
  Week 0, n = 183 | 5.76 (9.28)
  Week 4, n = 168 | 5.23 (0.97)
  Week 10, n = 168 | 7.53 (16.82)
  Week 16, n = 157 | 8.30 (37.90)

23. Secondary Outcome: Mean Serum Sodium Over Time
Description: Mean values of serum sodium are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MIRCERA
Number analyzed (Participants) | 184
mmol/L
  Week 0, n = 184 | 136.4 (10.67)
  Week 4, n = 168 | 136.3 (11.32)
  Week 10, n = 168 | 133.9 (20.98)
  Week 16, n = 156 | 137.0 (11.19)

24. Secondary Outcome: Mean Serum Phosphate Over Time
Description: Mean values of serum phosphate are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 166
mg/dL
  Week 0, n = 166 | 6.20 (7.50)
  Week 4, n = 156 | 6.32 (7.58)
  Week 10, n = 155 | 8.71 (34.13)
  Week 16, n = 146 | 6.17 (2.16)

25. Secondary Outcome: Mean Serum Bilirubin Over Time
Description: Mean values of serum bilirubin are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 142
mg/dL
  Week 0, n = 142 | 0.58 (0.32)
  Week 4, n = 124 | 0.68 (0.86)
  Week 10, n = 123 | 0.70 (1.08)
  Week 16, n = 117 | 0.62 (0.50)

26. Secondary Outcome: Mean Aspartate Transaminase Over Time
Description: Mean values of aspartate transaminase are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | MIRCERA
Number analyzed (Participants) | 184
Units/Liter (U/L)
  Week 0, n = 184 | 22.33 (13.06)
  Week 4, n = 171 | 21.69 (14.93)
  Week 10, n = 166 | 24.61 (19.44)
  Week 16, n = 157 | 22.63 (18.53)

27. Secondary Outcome: Mean Alanine Aminotransferase Over Time
Description: Mean values of alanine aminotransferase are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MIRCERA
Number analyzed (Participants) | 185
U/L
  Week 0, n = 185 | 27.89 (19.38)
  Week 4, n = 171 | 26.80 (21.57)
  Week 10, n = 166 | 28.11 (25.02)
  Week 16, n = 157 | 29.21 (24.45)

28. Secondary Outcome: Mean Serum Alkaline Phosphatase Over Time
Description: Mean values of serum alkaline phosphatase are presented at Baseline (Week 0), Week 4, Week 10, and Week 16.
Time Frame: Baseline (Week 0), Week 4, Week 10, and Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MIRCERA
Number analyzed (Participants) | 175
U/L
  Week 0, n = 175 | 176.2 (208.4)
  Week 4, n = 159 | 161.7 (197.8)
  Week 10, n = 156 | 161.7 (172.7)
  Week 16, n = 145 | 153.5 (135.2)

ADVERSE EVENTS:
Time Frame: Up to Week 18
Description: Safety population included all participants who receive at least one dose of study drug.
Arm/Group | MIRCERA
Serious Adverse Events (participants affected / at risk) | 24/189
Other Adverse Events (participants affected / at risk) | 11/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=189)
Cardio-respiratory arrest (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 4
Cellulitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Diabetic foot (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Amputation (Surgical and medical procedures) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 2
Accelerated hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=189)
Pyrexia (General disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.